CLINICAL TRIAL: NCT03452930
Title: A Phase I Study to Investigate the Safety, Pharmacokinetic Profile and the Efficacy of EDO-S101, a First-in-Class Alkylating HDACi Fusion Molecule in Patients With Newly Di-Agnosed MGMT-Promoter Unmethylated Glioblastoma
Brief Title: Tinostamustine With or Without Radiation Therapy in Treating Patients With Newly Diagnosed MGMT-Unmethylated Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0555; NCI-2018-00872 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0555 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-02-16; First posted 2018-03-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-06

CONDITIONS: Glioblastoma; Gliosarcoma; MGMT-Unmethylated Glioblastoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Radiotherapy; Radiation; tinostamustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stage 1 (tinostamustine) (Experimental): Patients who have completed TMZ and RT receive tinostamustine IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Tinostamustine
- Stage 2 (RT, tinostamustine) (Experimental): Patients who have received no treatment other than surgery undergo RT 5 days a week for up to 6 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive tinostamustine over 60 minutes IV on day 1. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiation Therapy; Drug: Tinostamustine

INTERVENTIONS:
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Stage 2 (RT, tinostamustine)
Drug: Tinostamustine — Given IV
  Other Names: 1H-Benzimidazole-2-heptanamide, 5-(Bis(2-chloroethyl)amino)-N-hydroxy-1-methyl-; EDO-S 101; EDO-S-101; EDO-S101

SUMMARY:
This phase I trial studies the side effects and best dose of tinostamustine (EDO-S101) given with or without radiation therapy in treating patients with newly diagnosed MGMT-unmethylated glioblastoma. Tinostamustine may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth in patients with glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the safety profile and determine the maximum tolerated dose (MTD) of tinostamustine (EDO-S101) in the adjuvant phase of therapy for patients with newly diagnosed MGMT-promoter unmethylated glioblastoma (GB) post chemoradiation with temozolomide. (Stage 1) II. To characterize the safety profile and determine the MTD of EDO-S101 when given as a single agent in the concomitant phase with radiation therapy (RT) in patients with newly diagnosed GB who are MGMT-promoter unmethylated. (Stage 2) III. To confirm the MTD of EDO-S101 in the concomitant phase and adjuvant phase in an expanded population of newly diagnosed GB patients who are MGMT-promoter un-methylated. (Dose Expansion Group)

SECONDARY OBJECTIVE:

I. To assess anti-tumor activity for patients with newly diagnosed GB who are MGMT-promoter unmethylated based on progression-free survival (PFS), overall survival (OS), and overall response rate (ORR).

EXPLORATORY OBJECTIVE:

I. Profiling tumor deoxyribonucleic acid (DNA), messenger ribonucleic acid (mRNA), microRNA and epigenetic profiling (DNA methylation) and evaluation of whole exome sequencing, RNA sequencing, microRNA sequencing and cell-free circulating tumor DNA (ctDNA) and correlate with outcome.

OUTLINE: This is a dose-escalation study of tinostamustine. Patients are assigned to 1 of 2 stages.

STAGE 1: Patients who have completed temozolomide (TMZ) and radiation therapy (RT) receive tinostamustine intravenously (IV) over 60 minutes on day 1. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

STAGE 2: Patients who have received no treatment other than surgery undergo RT 5 days a week for up to 6 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive tinostamustine over 60 minutes IV on day 1. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Have histologically confirmed World Health Organization grade IV glioma (glioblastoma [GB] or gliosarcoma).
* Patients must have preliminary glioblastoma (GBM) MGMT status (tumor must be MGMT promoter unmethylated) determined prior to study entry. If initial MGMT status is determined to be "unmethylated", by an outside institution the patient may be enrolled and begin treatment. However, MGMT status must be retested following enrollment by central laboratory Clinical Laboratory Improvement Act (CLIA) certified testing at MD Anderson, if tissue is available. Confirmed IDH wildtype. The presence of an IDH mutation will be an exclusionary criteria for trial enrollment.
* Have a performance status of >= 60 on the Karnofsky performance scale (KPS).
* If patient is on steroids, patient must be on a stable or decreasing dose of steroids for at least 5 days at the time of baseline brain magnetic resonance imaging (MRI).
* Absolute neutrophil count (ANC) >= 1,500 /mcL (within 14 days [+3 working days] of treatment initiation).
* Platelets >= 100,000 /mcL (within 14 days [+3 working days] of treatment initiation).
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (within 14 days [+3 working days] of treatment initiation).
* Serum creatinine OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) =< 1.5 x upper limit of normal (ULN) OR >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN (within 14 days [+3 working days] of treatment initiation).
* Serum total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (within 14 days [+3 working days] of treatment initiation).
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (within 14 days [+3 working days] of treatment initiation).
* International normalized ratio (INR) or prothrombin time (PT), activated partial thromboplastin time (aPTT) =< 1.5 x ULN (within 14 days [+3 working days] of treatment initiation).
* Female subjects of childbearing potential should have a negative serum pregnancy test within 72 hours of starting first dose of study drug.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the duration of the study. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception during the course of the study.
* Patients must have completed standard radiation therapy with concurrent TMZ and must not have evidence of progressive disease on post treatment imaging. Progression can only be defined using diagnostic imaging if there is new enhancement outside of the radiation field (beyond the high-dose region or 80% isodose line) or if there is unequivocal evidence of viable tumor on histopathologic sampling (e.g., solid tumor areas [i.e, > 70% tumor cell nuclei in areas], high or progressive increase in MIB-1 proliferation index compared with prior biopsy, or evidence for histologic progression or increased anaplasia in tumor). Note: Given the difficulty of differentiating true progression from pseudoprogression, clinical decline alone, in the absence of radiographic or histologic confirmation of progression, will not be sufficient for definition of progressive disease in the first 12 weeks after completion of concurrent chemoradiotherapy. (For Stage 1: post-chemoradiation group only)
* Prescribed treatment with concomitant temozolomide must be consistent with the Food and Drug Administration (FDA) package insert. The dose must be 75 mg/m^2 daily for the 6 to 6.5 weeks of radiation therapy. If the patient missed more than 1 week of temozolomide dosing during radiotherapy, then they are not eligible for the trial. EDO-S101 can accentuate thrombocytopenia induced by temozolomide. Therefore, if patients had a platelet < 75,000/mm^3 during concomitant temozolomide therapy during radiation, they are not eligible for this trial

  * NOTE: Complete blood count (CBC) should be monitored during chemoradiation and lowest platelet count must be submitted at registration. (For stage 1: post-chemoradiation group only)
* Patients must have undergone surgery of their GBM, and must not have had any further treatment following surgery. A minimal interval of 7 days between the day of surgery and the day of inclusion should be respected; a maximal interval of 31 days between the day of surgery and the day of inclusion should be respected; the patient should have fully clinically recovered from the surgery. (For stage 2: radiation with concurrent and adjuvant EDO-S101 only)
* Patients must undergo surgery and must not have further treatment. (For MTD expansion cohort only)

Exclusion Criteria:

* Has received prior interstitial brachytherapy, implanted chemotherapy, or therapeutics delivered by local injection or convection enhanced delivery. Prior treatment with Gliadel wafers will be excluded. Concomitant use of the Optune device will also be excluded.
* Is currently participating or has participated in any other any other investigational or therapeutic trial before or after chemoradiation.
* Any serious medical condition that interferes with adherence to study procedures.
* Has had prior chemotherapy, targeted small molecule therapy, within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent. Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy. (For Stage 1: post-chemoradiation group only)
* Patients with a history of a second malignancy diagnosed within three (3) years of study enrollment or have a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* New York Heart Association (NYHA) stage III/IV congestive heart failure, arrhythmias not adequately controlled.
* Patients with prolonged corrected QT (QT) interval defined as male > 450 msec and female > 470 msec.
* Patients who are on treatment with drugs known to prolong the QT/QTc interval. Case of the selective serotonin reuptake inhibitors (SSRIs): Patients treated with a SSRI AND displaying a QTc prolongation are NOT eligible in the trial. Nevertheless, there is no need to stop or change a SSRI if a patient is on a stable dose AND with no impact on QT/QTc interval, since it is not expected that plasma concentration of the SSRI will be affected by the administration of EDO-S101
* Serum potassium and magnesium within normal range, at baseline (supplementation is permissible)
* Has known gliomatous meningitis, extracranial disease, or multifocal disease. Subject has multifocal GBM, defined as discrete sites of contrast enhancing disease without contiguous T2/fluid-attenuated inversion recovery (FLAIR) abnormality that require distinct radiotherapy ports. Satellite lesions that are associated with a contiguous area of T2/FLAIR abnormality as the main lesion(s) and that are encompassed within the same radiotherapy port as the main lesion(s) are permitted.
* Has an active infection requiring systemic therapy.
* Has an ongoing or previous history of spontaneous intratumoral hemorrhage.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit.
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies). Testing not required.
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus (HCV) RNA [qualitative] is detected). (Testing not required for stage 2 and MTD expansion cohort)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Contraindication for undergoing MRIs.
* Use of any drug with histone deacetylase (HDAC) inhibiting activity.
* Use of valproate in any of its indications (epilepsy, mood disorder). Valproate, due to its HDAC inhibiting activity is contraindicated. For those patients on valproate, valproate will need to be discontinued and switched to a different anti-epileptic agent or psychotropic agent. A washout period of 4 days from valproate acid will be allowed prior to enrolling into the trial.
* Patients who missed more than 1 week of temozolomide dosing during radiotherapy. (For Stage 1: Post-chemoradiation group only)
* Patients who had a platelet < 75,000/mm^3 during concomitant temozolomide therapy during radiation. (For Stage 1: Post-chemoradiation group only)
* Has had any prior chemotherapy, targeted small molecule therapy. (For Stage 2: Radiation with concurrent and adjuvant EDO-S101 and MTD Expansion cohort only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Stages 1 & 2) | Up to 4 weeks
  Defined by dose limiting toxicity (DLT). Toxicity will be evaluated according to the most current version of the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) toxicity criteria. The MTD is confirmed when six (6) patients are treated at a dose level with less than two (2) DLTs.

SECONDARY OUTCOMES:
Incidence of adverse events (Stage 1) | Up to 2 years
  Graded according to CTCAE version 4.0. Toxicity monitoring will be conducted using Bayesian continuous monitoring, where the toxicity evaluation endpoint is defined as treatment-related unmanageable toxicities, including grade >= 3 AEs that require termination of the treatment during cycle one. Toxicity rate of 30% or higher will be considered unacceptable. The overall toxicity rate will be summarized by frequency and 95% confidence interval. Adverse Events will be tabulated by grade and by their relationship to the treatment.
Objective response rate (ORR) (Stage 2) | Up to 2 years
  The ORR will be summarized by frequency and 95% confidence interval. Logistic regression will be used to explore the correlation between response rates.
Overall survival (OS) (Stage 2) | Up to 2 years
  Kaplan-Meier curves will be generated and median survival time will be derived for OS. Cox proportional hazard regression will be employed for multivariate analysis on time-to-event outcomes with factors.
Progression-free survival (PFS) (Stage 2) | Up to 2 years
  Kaplan-Meier curves will be generated and median survival time will be derived for PFS. Cox proportional hazard regression will be employed for multivariate analysis on time-to-event outcomes with factors.

CONTACTS AND LOCATIONS:
Overall Officials: Shiao-Pei S Weathers, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org